CLINICAL TRIAL: NCT07114991
Title: Effects of Pedal-Assist E-Bike Commuting on Cardiometabolic Health, Physical Activity, and Psychological Well-Being in Overweight College Students
Brief Title: E-Bike Commuting and Health in Overweight College Students
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, River Falls (Other)
Responsible Party: Principal Investigator, Gregory Ruegsegger, Professor, University of Wisconsin, River Falls
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-101
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Obesity &Amp; Overweight; Sedentary Behaviors; Cardiometabolic Risk; Physical Inactivity
Keywords: Electric bicycle; Active commuting; Exercise motivation; Health behavior; Physical activity; Overweight
MeSH Terms: conditions — Obesity; Overweight; Sedentary Behavior; Health Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants in this group will receive a pedal-assist electric bicycle (e-bike), helmet, safety training, and cycling computer. They will be instructed to use the e-bike for commuting or transportation at least four days per week for 12 weeks. They will also complete assessments at baseline, Week 12, and Week 24, including fitness testing, body composition, blood testing, surveys, and activity monitoring.
  Interventions: Behavioral: E-Bike Commuting
- Control Group (No Intervention): Participants in the control group will maintain their usual commuting and physical activity habits for the 12-week intervention period. They will complete the same assessments as the intervention group at baseline, Week 12, and Week 24.

INTERVENTIONS:
Behavioral: E-Bike Commuting — Participants in the intervention group will receive a pedal-assist electric bicycle (e-bike), a helmet, safety training, and a cycling computer. They will be asked to use the e-bike for commuting or personal travel at least four times per week for 12 weeks. E-bike usage will be monitored using a Garmin Edge device. Participants will also complete baseline, 12-week, and 24-week assessments including fitness testing, blood tests, body composition, surveys, and wearable activity monitoring.
  Arms: Experimental Group

SUMMARY:
This study will evaluate the effects of using a pedal-assist electric bicycle (e-bike) for commuting on physical activity, fitness, and health in overweight or obese college students. Participants will be randomly assigned to either a 12-week e-bike commuting intervention or a control group. The study will measure changes in cardiorespiratory fitness, body composition, blood biomarkers, physical activity, and psychological well-being over a 24-week period.

DETAILED DESCRIPTION:
This randomized controlled trial investigates the effectiveness of e-bike commuting as a strategy to improve cardiometabolic health, physical activity levels, and psychological well-being in college students with a body mass index (BMI) of 25 kg/m² or higher. Eligible participants will be randomized to either a 12-week e-bike intervention group or a control group that continues usual commuting habits. Assessments will occur at baseline (Week 0), post-intervention (Week 12), and follow-up (Week 24). Each assessment will include VO₂peak testing using a graded cycle ergometer protocol, body composition assessment via BodPod, fasting fingerstick blood tests for glucose, cholesterol, and triglycerides, blood pressure and resting heart rate measurement, and self-report questionnaires evaluating motivation, stress, affect, mental health, and academic engagement. Participants will also complete a 30-minute submaximal cycling test during which affective responses will be recorded, and physical activity will be tracked over 7 days. Those assigned to the intervention group will receive a pedal-assist e-bike, helmet, and safety training and will be asked to ride at least four days per week for 12 weeks. The study aims to determine whether e-bike commuting can promote sustained physical activity and improve cardiometabolic and mental health outcomes in a population at risk for early health decline.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-29 years
* Currently enrolled undergraduate or graduate student
* Body mass index (BMI) ≥25.0 kg/m² (classified as overweight or obese)
* Self-report of engaging in <150 minutes per week of moderate-to-vigorous physical activity
* Able and willing to safely ride a bicycle for commuting or transportation purposes
* Willing to be randomized and complete all study procedures across 24 weeks Able to provide informed consent

Exclusion Criteria:

* Current use of a bicycle or e-bike for commuting ≥2 times per week
* Known cardiovascular, metabolic, or orthopedic conditions that limit physical activity or make exercise testing unsafe
* Currently pregnant, planning pregnancy during the study period, or less than 6 months postpartum
* Use of medications known to affect glucose metabolism, heart rate, or physical activity (e.g., beta-blockers, insulin)
* Diagnosed severe mental health disorders that would impair study participation
* Participation in another clinical trial or lifestyle intervention within the past 3 months
* Inability or unwillingness to attend lab visits or comply with the intervention protocol

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in daily moderate-to-vigorous physical activity (minutes/day) | From enrollment to end of study at 24 weeks.
  Physical activity will be measured using a hip-worn ActiGraph GT3X+ accelerometer over 7 consecutive days at baseline, Week 12, and Week 24. The device will be analyzed using validated cut points to determine average daily time spent in moderate-to-vigorous physical activity (MVPA). The primary outcome is the change in MVPA from baseline to Week 24
Change in cardiorespiratory fitness (VO₂peak, mL/kg/min) | From enrollment to end of study at 24 weeks.
  Cardiorespiratory fitness will be measured via a graded cycling test using a metabolic cart to determine peak oxygen uptake (VO₂peak). Participants will complete the test at baseline (Week 0), post-intervention (Week 12), and follow-up (Week 24). The primary comparison will be the change in VO₂peak from baseline to Week 12 between the intervention and control groups.

SECONDARY OUTCOMES:
Change in body fat percentage | From enrollment to end of study at 24 weeks.
  Body composition will be assessed using air displacement plethysmography (BodPod®). Percent body fat will be calculated at baseline, Week 12, and Week 24.
Change in total cholesterol, HDL-C, LDL-C, and triglycerides (mg/dL) | From enrollment to end of study at 24 weeks.
  Fasting lipid profiles will be assessed at baseline, Week 12, and Week 24 via fingerstick blood sample. Changes in total cholesterol, HDL, LDL, and triglycerides will be evaluated to assess cardiometabolic risk.
Change in fasting blood glucose (mg/dL) | From enrollment to end of study at 24 weeks.
  Fasting blood glucose will be collected via fingerstick and analyzed using a portable blood analyzer. Values will be compared between baseline, Week 12, and Week 24 to determine the impact of the e-bike intervention on glucose regulation.
Change in exercise motivation (BREQ-3 score) | From enrollment to end of study at 24 weeks.
  Exercise motivation will be assessed using the Behavioral Regulation in Exercise Questionnaire-3 (BREQ-3) at all three time points. Subscale scores (e.g., intrinsic motivation, external regulation) will be analyzed for changes between baseline, Week 12, and Week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Ruegsegger, PhD, Principal Investigator — University of Wisconsin, River Falls
Locations (1):
- University of Wisconsin-River Falls, River Falls, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) collected in this study-including demographic information, outcome measures (e.g., physical activity, VO₂peak, body composition, survey scores), and visit-level data-will be made available to qualified researchers upon reasonable request. Data will be shared in a manner that protects participant confidentiality and complies with IRB and institutional policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 12 months after study completion and for up to 5 years thereafter.
Access Criteria: Researchers must submit a data use request, including a brief study proposal and data security plan, to the study principal investigator. Requests will be reviewed by the research team for scientific merit and feasibility. Approved researchers will be provided with a de-identified dataset via a secure, password-protected data repository.

REFERENCES:
- [Background] Peterman JE, Morris KL, Kram R, Byrnes WC. Pedelecs as a physically active transportation mode. Eur J Appl Physiol. 2016 Aug;116(8):1565-73. doi: 10.1007/s00421-016-3408-9. Epub 2016 Jun 14. PMID 27299435
- [Background] Berntsen S, Malnes L, Langaker A, Bere E. Physical activity when riding an electric assisted bicycle. Int J Behav Nutr Phys Act. 2017 Apr 26;14(1):55. doi: 10.1186/s12966-017-0513-z. PMID 28446180
- [Background] Johnson L, O'Hara BJ, Phongsavan P, et al. Exploring the feasibility of a 6-week electric-bike intervention with behavioural support in Australia. International Journal of Environmental Research and Public Health. 2021;18(16):8684
- [Background] Bourne JE, Sauchelli S, Perry R, Page A, Leary S, England C, Cooper AR. Health benefits of electrically-assisted cycling: a systematic review. Int J Behav Nutr Phys Act. 2018 Nov 21;15(1):116. doi: 10.1186/s12966-018-0751-8. PMID 30463581